CLINICAL TRIAL: NCT02689102
Title: Confocal Laser Endomicroscopy and OCT for Diagnosing ILD, a Comparison With Imaging and Pathology.
Brief Title: Confocal Laser Endomicroscopy and Optical Coherence Tomography for Diagnosing ILD.
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Prof J.T. Annema, prof.dr. J.T. Annema, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: NL 54612.018.15
Record Dates: First submitted 2016-01-28; First posted 2016-02-23 (Estimated); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: Interstitial Lung Diseases
Keywords: Optical coherence tomography; Confocal laser endomicroscopy
MeSH Terms: conditions — Lung Diseases, Interstitial | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ILD patients: ILD patients scheduled for diagnostic bronchoscopy with biopsy and/or broncho-alveolar lavage will undergo additional imagaing with probe based optical techniques.
  Interventions: Device: Probe based optical techniques

INTERVENTIONS:
Device: Probe based optical techniques — During the diagnostic bronchoscopy, optical biopsy of the mucosa and alveolar compartment will be conducted by two different probe based optical techniques (Confocal Laser Endomicroscopy (Mauna Kea technologies) and Optical Coherence Tomography (St Jude Medical)). After the study measurements a biopsy will be obtained in the same area.
  Other Names: Confocal Laser Endomicroscopy (Mauna Kea technologies); Optical Coherence Tomography (St Jude medical)

SUMMARY:
Often, assessing a classifying diagnosis in patients with interstitial lung disease provides a diagnostic challenge. Currently HRCT, endoscopic or surgical video assisted thoracoscopic surgery(VATS) assessment including lung biopsies are diagnostic tools for patients with suspected ILD. However, tissue acquisition is associated with morbidity in these patients with an already compromised pulmonary function. In clinical practice this results in the fact that only a minor part of patients with an indication for tissue acquisition are actually undergoing biopsies. The aim of this study is to determine ILD-characteristics on imagign collected with minimal invasive novel optical techniques, to examine whether the addition of novel optical techniques to the diagnostic process of ILD could potentially limit the need for a tissue- (surgical) diagnosis and/or reduce the sampling error rate of biopsies by providing additional information on biopsy location.

DETAILED DESCRIPTION:
Novel probe based optical techniques such as Confocal laser endomicroscopy (pCLE) and Optical coherence tomography (pOCT) are non-invasive optical techniques, compatible with conventional diagnostic bronchoscopes and provide non-invasive, real-time information on the airway wall and the alveolar compartment. Therefore, immediate validation of optical measurements during a biopsy is possible. Optical techniques might either obviate the need for an tissue biopsy or improve the diagnostic yield of conventional biopsy methods and make surgical lung biopsies that are associated with high morbidity and costs redundant.

Hypothesis: Novel optical techniques (pCLE and pOCT) provide real time information about the characteristics of the mucosa and/or the alveolar compartment in ILD.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age

  * Supected ILD and referred for diagnostic bronchoscopic procedure with cryobiopsy

Exclusion Criteria:

* Smoked in the last 6 months
* Inability and willingness to provide informed consent
* Inability to comply with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of 18 years or older (n=20), who are suspected for ILD based on imaging (HRCT-scan) and with an indication for bronchoscopy with cryobiopsy.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-10-28 (Actual); Primary Completion 2017-04-22 (Actual); Study Completion 2017-04-22 (Actual)

PRIMARY OUTCOMES:
Describing visual characteristics on CLE-imaging and pOCT imaging of ILD. | cross sectional (1 day)

SECONDARY OUTCOMES:
(um), size of the alveolar openings, number of cells on CLE imaging of the alveolar space (um). | cross-sectional (1 day)
Size of the alveolar openings (um), thickness of the alveolar septum/alveolar openings on pOCT imaging of the alveolar compartment (um). | cross-sectional (1day)
Feasibility of pOCT alveolar compartment: measuring number of alveoli, trajectory in OCT pull-back with alveoli (mm), number of study-related adverse events. | cross-sectional (1 day)
Correlation between pOCT imaging and histology (alveolar septum-thickness and alveolar space (um)) | cross-sectional (1 day)
Correlation between pOCT imaging and histology (alveolar septum thickness (um) and alveolar compartment (mm) | cross-sectional (1 day)

CONTACTS AND LOCATIONS:
Overall Officials: Jouke T Annema, MD, PhD, Principal Investigator — Netherlands, Academisch Medisch Centrum
Locations (1):
- Academisch Medisch Centrum, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
CLE and OCT imaging